CLINICAL TRIAL: NCT05719298
Title: Infant Respiratory Interface and Accessories Evaluation Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fisher and Paykel Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: UT-1111-1267-0940; CIA-235 (Other: Fisher & Paykel Healthcare)
Record Dates: First submitted 2023-01-31; First posted 2023-02-08 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-01

CONDITIONS: Respiratory Distress Syndrome, Newborn
MeSH Terms: conditions — Respiratory Distress Syndrome, Newborn

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Respiratory interface (Experimental): Use of the new respiratory interface and accessories to deliver non-invasive therapy
  Interventions: Device: Respiratory interface

INTERVENTIONS:
Device: Respiratory interface — Application of the new interface and accessories and provision of non-invasive respiratory support through the device.

SUMMARY:
Determine the usability of an interface and its accessories to provide non-invasive respiratory therapy to neonates and infants.

ELIGIBILITY:
Inclusion Criteria:

* Spontaneously breathing infants who require non-invasive respiratory support
* Parent(s)/guardian(s) at least 18 years of age

Exclusion Criteria:

* Parent(s)/guardian(s) unable to give written informed consent
* Neonate or infant not requiring non-invasive support
* Suspected or confirmed abnormalities or trauma to the skull or airway

Max Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Estimated)
Dates: Start 2023-02 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Feedback score | 12 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Mater Mothers' Hospital NICU, Brisbane, Queensland, Australia